CLINICAL TRIAL: NCT01308190
Title: Prospective Randomized Clinical Trial for no Inferiority With Preoperative Chemoradiotherapy and Transanal Endoscopic Microsurgery (TEM) Versus Total Mesorectal Excision in T2-T3s N0, M0 Rectal Cancer
Brief Title: Preoperative Chemoradiotherapy and Transanal Endoscopic Microsurgery Versus Total Mesorectal Excision in T2-T3s N0, M0 Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Fundación Olga Torres (Unknown)
Responsible Party: Principal Investigator, Xavier Serra-Aracil, Medical Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAU-TEM-2009-01
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Rectal Cancer
Keywords: Preoperative chemoradiotherapy; Transanal endoscopic microsurgery; Rectal Cancer; T2-T3s-N0
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Transanal Endoscopic Microsurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemoradiotherapy+TEM (Active Comparator): Preoperative chemotherapy: capecitabine 825 mg/m2 every 12 hours orally, plus Radiotherapy (50.4 Gy). After 6-8 weeks, transanal endoscopic microsurgery (TEM)is done
  Interventions: Drug: Capecitabine (Xeloda); Radiation: 50.4 Gy; Procedure: Transanal Endoscopic Microsurgery
- Total Mesorectal Excision (Other): Standard surgical treatment of T2 , T3s, N0, M0 rectal cancer
  Interventions: Procedure: Total Mesorectal Excision

INTERVENTIONS:
Drug: Capecitabine (Xeloda) — Capecitabine 825 mg/m2 every 12 hours orally on days of radiotherapy
  Arms: Chemoradiotherapy+TEM
Radiation: 50.4 Gy — Radiotherapy was administered in daily fractions of 1.8 Gy 5 days a week according to standard schema. The total dose is 45 Gy plus a boost of 5.4 Gy to the tumor area
  Arms: Chemoradiotherapy+TEM
Procedure: Transanal Endoscopic Microsurgery — 6-8 weeks after Chemoradiotherapy
  Arms: Chemoradiotherapy+TEM
Procedure: Total Mesorectal Excision — Standard surgical treatment of T2 , T3s, N0, M0 rectal cancer. Early after diagnosis
  Arms: Total Mesorectal Excision

SUMMARY:
The standard treatment of rectal adenocarcinoma is total mesorectal excision (TME). The technique involves a low anterior rectal or colo-anal resection, very often associated with a protective stoma or abdominal-perineal resection with permanent colostomy. Transanal endoscopic microsurgery (TEM) allows access to tumors up to 20 cm from the anal margin, with minimal postoperative morbidity and mortality. Recent studies of T1 rectal adenocarcinomas consider TEM to be the technique of choice. However the treatment of T2 rectal cancers remains controversial. Chemotherapy and radiotherapy (CT/RT) has achieved a concomitant reduction in local recurrence and an increase in survival.

Hypothesis: Patients with rectal adenocarcinoma less than 10 cm from the anal margin and up to 4 cm in size, staged after endorectal ultrasound and MRI as T2 or superficial T3 N0-M0-N0-M0, who underwent surgery after preoperative local chemoradiotherapy (TEM), achieve effective results in terms of local recurrence similar to radical surgery (TME).

OBJECTIVES:

Primary: To compare the results of local recurrence at 2 years in patients treated with preoperative chemoradiotherapy and TEM and in patients treated with conventional radical surgery (TME).

Secondary: To analyse the 3-year survival results in patients treated with CT/RT.

Methodology: Multicenter clinical trial in a calculated sample of 173 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Rectal adenocarcinomas located 10 cm or less from the inferior anal verge measured using a rigid rectoscope at the time of the EUS.
2. Preoperative staging by EUS and pelvic MRI of T2 or T3 superficial, N0. In case of disparity, the higher staging is considered as the definitive diagnosis.
3. Tumours equal to or less than 4 cm of diameter maximum measured using colonoscopy, EUS or MRI. We use the highest score on both scores.
4. ASA score III or less.
5. Absence of distance metastasis as shown on abdominal CT.

Exclusion Criteria:

1. Preoperative staging by EUS or pelvic MRI of T1, deep T3, T4 or N1.
2. Presence of distance metastasis.
3. Synchrony with other colorectal adenocarcinomas.
4. Undifferentiated rectal adenocarcinomas or with presence of poor prognosis factors in preoperative biopsy.
5. Patients with intolerance of preoperative chemotherapy or radiotherapy.
6. Refusal to sign informed consent to enter the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Local recurrence | 2 years
  To analyse the results for local recurrence after 2 years in patients treated with preoperative chemoradiotherapy and TEO, with patients treated with conventional radical surgery (TME).

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Background] Serra Aracil X, Bombardo Junca J, Mora Lopez L, Alcantara Moral M, Ayguavives Garnica I, Darnell Marti A, Casalots Casado A, Pericay Pijaume C, Campo Fernandez de Los Rios R, Navarro Soto S. [Site of local surgery in adenocarcinoma of the rectum T2N0M0]. Cir Esp. 2009 Feb;85(2):103-9. doi: 10.1016/j.ciresp.2008.09.007. Epub 2009 Feb 5. Spanish. PMID 19231466
- [Background] Serra-Aracil X, Vallverdu H, Bombardo-Junca J, Pericay-Pijaume C, Urgelles-Bosch J, Navarro-Soto S. Long-term follow-up of local rectal cancer surgery by transanal endoscopic microsurgery. World J Surg. 2008 Jun;32(6):1162-7. doi: 10.1007/s00268-008-9512-1. PMID 18338206
- [Derived] Serra-Aracil X, Pericay C, Cidoncha A, Badia-Closa J, Golda T, Kreisler E, Hernandez P, Targarona E, Borda-Arrizabalaga N, Reina A, Delgado S, Espin-Bassany E, Caro-Tarrago A, Gallego-Plazas J, Pascual M, Alvarez-Laso C, Guadalajara-Labajo H, Otero A, Biondo S; TAUTEM Collaborative Group. Chemoradiotherapy and Local Excision vs Total Mesorectal Excision in T2-T3ab, N0, M0 Rectal Cancer: The TAUTEM Randomized Clinical Trial. JAMA Surg. 2025 Jul 1;160(7):783-793. doi: 10.1001/jamasurg.2025.1398. PMID 40434784
- [Derived] Motamedi MAK, Mak NT, Brown CJ, Raval MJ, Karimuddin AA, Giustini D, Phang PT. Local versus radical surgery for early rectal cancer with or without neoadjuvant or adjuvant therapy. Cochrane Database Syst Rev. 2023 Jun 13;6(6):CD002198. doi: 10.1002/14651858.CD002198.pub3. PMID 37310167
- [Derived] Serra-Aracil X, Pericay C, Badia-Closa J, Golda T, Biondo S, Hernandez P, Targarona E, Borda-Arrizabalaga N, Reina A, Delgado S, Vallribera F, Caro A, Gallego-Plazas J, Pascual M, Alvarez-Laso C, Guadalajara-Labajo HG, Mora-Lopez L. Short-term outcomes of chemoradiotherapy and local excision versus total mesorectal excision in T2-T3ab,N0,M0 rectal cancer: a multicentre randomised, controlled, phase III trial (the TAU-TEM study). Ann Oncol. 2023 Jan;34(1):78-90. doi: 10.1016/j.annonc.2022.09.160. Epub 2022 Oct 8. PMID 36220461
- [Derived] Serra-Aracil X, Pericay C, Golda T, Mora L, Targarona E, Delgado S, Reina A, Vallribera F, Enriquez-Navascues JM, Serra-Pla S, Garcia-Pacheco JC; TAU-TEM study group. Non-inferiority multicenter prospective randomized controlled study of rectal cancer T2-T3s (superficial) N0, M0 undergoing neoadjuvant treatment and local excision (TEM) vs total mesorectal excision (TME). Int J Colorectal Dis. 2018 Feb;33(2):241-249. doi: 10.1007/s00384-017-2942-1. Epub 2017 Dec 12. PMID 29234923